CLINICAL TRIAL: NCT02457871
Title: Promoting Self-Management in Low Income African Americans Living With Hypertension
Acronym: ENCM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bev Zabler (Other)
Collaborators: Medical College of Wisconsin (Other)
Responsible Party: Sponsor-Investigator, Bev Zabler, Clinical Assistant Professor, University of Wisconsin, Milwaukee
Organization: University of Wisconsin, Milwaukee (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 144-PRJ94IR
Record Dates: First submitted 2015-05-28; First posted 2015-05-29 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2016-05

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ecological Nurse Case Managemnt (Experimental): Ecological Nurse Case Management (ENCM) group receives 6 months of ENCM services in addition to their usual primary care services at the study site.
  Interventions: Behavioral: Ecological Nurse Case Management
- Comparison (No Intervention): Usual Clinical Care - is the usual primary care services delivered at the site of the study, a free clinic.

INTERVENTIONS:
Behavioral: Ecological Nurse Case Management — The Ecological Nurse Case Management (ENCM) intervention allows for individualized case management based on client preferences through mutual goal setting and client choice points, nursing assessments, the nurse's analytic decision-making process and critical thinking, and nursing actions.
  Arms: Ecological Nurse Case Managemnt

SUMMARY:
The specific study aims are to: 1) examine differences between an Ecological Nursing Case Management (ENCM) treated group and a comparison group on self-efficacy, SM behaviors, and health status to establish effect sizes needed for a future large randomized controlled trial; 2) explore the dose-response of specific elements of the ENCM intervention; and 3) examine moderating effects of gender and perceived stress on the intervention effect. This is a two-group randomized experimental study with repeated measurements. Clients in the treatment group (n=25) will receive the individualized ENCM and those in the comparison group (n=25) will receive usual clinic care. Data will be collected at baseline, 1, 3, and 6 months to capture the immediate, short and longer term effects of the intervention.

DETAILED DESCRIPTION:
Health outcomes of chronically ill low-income adults are costly in both fiscal and human terms. Although advances have been made in understanding how nurse case management (NCM) can contribute to self-management (SM) behaviors, the factors that contribute to sustained SM behaviors in low-income African American populations are not well understood. This study will examine the impact of Ecological Nurse Case Management (ENCM) on self-management behaviors, health status, and self-efficacy of poor, chronically ill, African American adults. In addition, we will explore moderating effects to determine if the ENCM intervention is differentially effective based on gender or perceived stress. The study will use the UWM Automated Community Health Information System, a relational electronic health record, to document the individualized ECNM intervention and dose of the intervention. The specific study aims are to: 1) examine differences between an ENCM treated group and a comparison group on self-efficacy, SM behaviors, and health status to establish effect sizes needed for a future large randomized controlled trial; 2) explore the dose-response of specific elements of the ENCM intervention; and 3) examine moderating effects of gender and perceived stress on the intervention effect. This is a two-group randomized experimental study with repeated measurements. Clients in the treatment group (n=25) will receive the individualized ENCM and those in the comparison group (n=25) will receive usual clinic care. Data will be collected at baseline, 1, 3, and 6 months to capture the immediate, short and longer term effects of the intervention. Acknowledging the small sample size, mixed models for repeated measures data (at baseline and M1, 3, and 6 post-intervention) will be fit to interactions involving moderating variables of gender and stress. The ENCM intervention draws on evidence that given the proper tools (i.e., knowledge, skills and support), individuals can learn to better self-manage their symptoms on a day to day basis and better utilize the health care resources available to them.

ELIGIBILITY:
Inclusion Criteria:

* Hypertension diagnosis Attend Bread of Healing Clinic

Exclusion Criteria:

* No Hypertension diagnosis Do not Attend Bread of Healing Clinic

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2014-07; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Change measures | @ baseline,one month, three months, six months
  NIH Toolbox Perceived Stress Survey NIH Toolbox Self-efficacy Survey Hypertension Self-Care Profile Blood pressure, BMI and Waist Circumference changes Hypertension Self-Care Profile

SECONDARY OUTCOMES:
Automated Community Health Information System (ACHIS) data elements | 6 months
  Data elements of ACHIS, including Omaha System informatics codes, will be used to measure the intervention dose and intervention outcomes of nurse rated knowledge and client self-reported health status.

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Schiffman, Ph.D., Study Director — University of Wisconsin-Milwaukee College of Nursing
Locations (1):
- University of Wisconsin Milwaukee College of Nursing, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No